CLINICAL TRIAL: NCT02162836
Title: A Phase 1 Study of Androgen Receptor (AR) Antagonist JNJ-56021927 in Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Safety Study of JNJ-56021927 in Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR103653; 56021927PCR1008 (Other: Janssen Pharmaceutical K.K)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: Prostatic Neoplasms, Castration-Resistant; Metastatic Castration-Resistant Prostate Cancer; Prostate Cancer; Androgen Receptor; JNJ-56021927
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms; Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Participants will receive 8 capsules of JNJ-56021927, 240 milligram (mg) as single oral dose on Day 1. After participants will receive daily JNJ-56021927, 240 mg on Day 1 of Cycle 1 until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first.
  Interventions: Drug: JNJ-56021927

INTERVENTIONS:
Drug: JNJ-56021927 — Participants will receive 8 capsules of JNJ-56021927, 240 milligram (mg) as single oral dose on Day 1. After participants will receive daily JNJ-56021927, 240 mg on Day 1 of Cycle 1 until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of JNJ-56021927 in Japanese participants with metastatic castration-resistant prostate cancer (mCRPC- prostate cancer that is resistant to medical [for example. hormonal] or surgical treatments).

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label (participants will know the identity of study drug received) study in participants with Metastatic Castration-Resistant Prostate Cancer (mCRPC). The study consists of 4 parts: Screening (28 days before study commences on Day 1), pharmacokinetic week (PK), Continuous daily dosing, Extension and Safety follow-up period. In PK week participants will receive a single oral capsule of JNJ-56021927 at a dose of 240 milligram (mg) on Day 1 and will be monitored for 1 week. After Week 1, in continuous daily dosing period, participants will receive continuous daily therapy at the same dose for 4 weeks (Cycle 1). After Cycle 1 participants, who will not meet the criteria for discontinuation listed such as progressive disease (PD) or unacceptable toxicity, will continue in safety follow-up period and will receive continuous daily therapy at the same dose up to cycle 13. Primarily dose limiting toxicity (DLT) will be evaluated. Participants' safety will be monitored throughout.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features, with metastatic disease
* Castration-resistant prostate cancer (CRPC) demonstrated during continuous androgen deprivation therapy (ADT)/post orchiectomy
* Maintain castrate levels of testosterone (less than [<] 50 nanogram per deciliter (ng/dL) [1.72 nanomol per liter {nmol/L}]) within 4 weeks before enrollment
* Prostate-specific antigen (PSA) evidence for progressive prostate cancer consists of a PSA level of at least greater than or equal to (>=) 2 nanogram per milliliter (ng/mL) within 2 weeks before enrollment which has risen on at least 2 successive occasions, at least 1 week apart. If the confirmatory PSA value is less than the last PSA value, then an additional test for rising PSA will be required to document progression
* Participants who received a first generation anti-androgen [for example, bicalutamide, flutamide, nilutamide (not approved in Japan)] as part of an initial combined androgen blockade therapy or as second-line hormonal therapy must show continuing disease progression off the anti-androgen for at least 4 weeks prior to the first dose of study drug

Exclusion Criteria:

* History of, or current metastases in the brain or untreated spinal cord compression
* Participants with progressive epidural disease
* Participants has a history of another malignancy within 5 years before screening
* Prior treatment with second generation anti-androgens ( for example, enzalutamide) or Cytochrome P450 17 (CYP 17) inhibitors [for example, abiraterone acetate, orteronel, galeterone, systemic ketoconazole (not approved in Japan, respectively)]
* Participants had used radiopharmaceutical agents (for example, Strontium-89) or investigational immunotherapy (for example, sipuleucel-T) within 12 weeks before the first dose of study drug

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicity | Week 1 up to Day 28 of Cycle 1
  The dose will be considered intolerable if a participants developed either any Grade 3 or 4 non-hematologic toxicity; GI toxicities such as abdominal pain, nausea, vomiting, constipation, and diarrhea, must persist at Grade 3-4 despite maximal medical therapy, Grade 4 neutropenia (that is, ANC less than [<] 500 per microliter [mcL] for five or more consecutive days, Grade 4 thrombocytopenia (<25,000 per mcL) or Grade 3 thrombocytopenia (greater than or equal to [>=] 25,000 - <50,000 per mcL) with a bleeding episode requiring platelet transfusion, any other Grade 4 hematologic toxicity of more than 5 days duration, any grade treatment-related seizure, the other toxicities which do not meet any of the above criteria but which, in the opinion of the Investigator, are equivalent to DLTs.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (C[max]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 and 96 hours post administration of study drug
  The C(max) is the maximum plasma concentration which will be observed at the defined time points.
Time to Reach the Maximum Plasma Concentration (T[max]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 and 96 hours post administration of study drug
  The T[max] is time to reach the observed maximum plasma concentration.
Elimination Half-life (t1/2[lambda]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 and 96 hours post administration of study drug
  Elimination half-life associated with the terminal slope (lambda[z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda (z).
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 and 96 hours post administration of study drug
  The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-last]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 and 96 hours post administration of study drug
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero time of the last quantifiable concentration C(last), and C(last) is the last observed quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 and 96 hours post administration of study drug
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z), wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Change in Prostate-specific Antigen (PSA) | Baseline, Day 1 of each cycle (28 days) until disease progression and up to 28 days after the last dose study drug
  Change in prostate specific antigen will be assessed using the Prostate Cancer Working Group 2 (PCWG2) criteria and Response Criteria in Solid Tumors (RECIST). PSA progression will delayed if decline from baseline: greater than or equal to (>=) 25 percent (%) and >= 2 nanogram per milliliter (ng/mL) above the PSA nadir, which is confirmed by a second value 3 or more weeks later; and no decline from baseline: PSA progression >= 25% and >= 2 ng/mL after 12 weeks.
Trough Plasma Concentration (C[trough]) | Pre- dose on Day 1 of Cycle 2 up to Cycle 13
  Trough plasma concentration (C[trough]) just before dosing will be assessed.
Observed Accumulation Index (A[cc] Index) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 and 96 hours post administration of study drug in Cycle 1
  Observed Accumulation Index (A[cc] Index) will be calculated as AUC[0-24] at steady state divided by AUC[0-24].
Effective Half-life (EHL) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 and 96 hours post administration of study drug in Cycle 1
  Effective Half-life (EHL) will be calculated as dosing interval minus log 2 divided by log {1-[1/A[cc]Index}.
Percent Peak to Trough Fluctuation (PTF) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 and 96 hours post administration of study drug in Cycle 1
  Percent Peak to Trough Fluctuation (PTF) will be calculated as 100 multiplied by {C[max]/C[min]}.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trials, Study Director — Janssen Pharmaceutical K.K.
Locations (4):
- Japan (4):
  - Fukuoka
  - Gifu
  - Matsuyama
  - Yokohama

REFERENCES:
- [Result] Tsuchiya T, Imanaka K, Iwaki Y, Oyama R, Hashine K, Yamaguchi A, Uemura H. An open-label, phase 1 study of androgen receptor antagonist, apalutamide in Japanese patients with metastatic castration-resistant prostate cancer. Int J Clin Oncol. 2019 Dec;24(12):1596-1604. doi: 10.1007/s10147-019-01526-7. Epub 2019 Aug 24. PMID 31446511
- [Derived] Uemura H, Koroki Y, Iwaki Y, Imanaka K, Kambara T, Lopez-Gitlitz A, Smith A, Uemura H. Skin rash following Administration of Apalutamide in Japanese patients with Advanced Prostate Cancer: an integrated analysis of the phase 3 SPARTAN and TITAN studies and a phase 1 open-label study. BMC Urol. 2020 Sep 2;20(1):139. doi: 10.1186/s12894-020-00689-0. PMID 32878613